CLINICAL TRIAL: NCT01979744
Title: Intravascular ULTrasound Guided Versus Conventional Angiography Guided Strategy to Deploy Zotarolimus and Everolimus Eluting Third Generation Stents in the Long Coronary Artery Lesions: ULTRA-ZET Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2013-0052
Record Dates: First submitted 2013-10-24; First posted 2013-11-08 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease
Keywords: Intravenous ultrasound,; third generation drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Resolute Integrity - IVUS (Experimental): Resolute Integrity - IVUS arm
  Interventions: Procedure: IVUS guided percutaneous coronary angioplasty with Resolute integrity stent insertion
- Resolute Integrity - Angio (Active Comparator): Resolute Integrity - Angio arm
  Interventions: Device: Angiography guided percutaneous coronary angioplasty with Resolute integrity stent insertion
- Promus - Angio (Active Comparator): Promus - Angio arm
  Interventions: Device: Angiography guided percutaneous coronary angioplasty with Promus element stent implantation
- Promus - IVUS (Active Comparator): Promus - IVUS arm
  Interventions: Procedure: Angiography guided percutaneous coronary angioplasty with Promus element stent implantation

INTERVENTIONS:
Procedure: IVUS guided percutaneous coronary angioplasty with Resolute integrity stent insertion — Resolute integrity stent implantation (diameter from 2.5mm to 3.5mm, length 30, 34, 38mm) The size and number of stents and post-dilation will be determined on physician's discrete within the range allowed in this study protocol. All procedure will be performed according to current standard technique. IVUS will be used to assess the anatomic characteristics of lesion and determine appropriate stent size and length. Additional stent implantation or post dilation will be allowed according to attending physician's discrete based on IVUS results.
  Arms: Resolute Integrity - IVUS
Device: Angiography guided percutaneous coronary angioplasty with Resolute integrity stent insertion — Resolute integrity stent implantation (diameter from 2.5mm to 3.5mm, length 30, 34, 38mm) The size and number of stents and post-dilation will be determined on physician's discrete within the range allowed in this study protocol. All procedure will be performed according to current standard technique. Additional stent implantation or post dilation will be allowed according to attending physician's discrete. IVUS will be not used in this arm.
  Arms: Resolute Integrity - Angio
Device: Angiography guided percutaneous coronary angioplasty with Promus element stent implantation — Promus element stent implantation (diameter from 2.5mm to 3.5mm, length 28, 32, 36mm) The size and number of stents and post-dilation will be determined on physician's discrete within the range allowed in this study protocol. All procedure will be performed according to current standard technique. Additional stent implantation or post dilation will be allowed according to attending physician's discrete. IVUS will be not used in this arm.
  Arms: Promus - Angio
Procedure: Angiography guided percutaneous coronary angioplasty with Promus element stent implantation — Promus element stent implantation (diameter from 2.5mm to 3.5mm, length 28, 32, 36mm) The size and number of stents and post-dilation will be determined on physician's discrete within the range allowed in this study protocol. All procedure will be performed according to current standard technique. IVUS will be used to assess the anatomic characteristics of lesion and determine appropriate stent size and length. Additional stent implantation or post dilation will be allowed according to attending physician's discrete based on IVUS results.
  Arms: Promus - IVUS

SUMMARY:
Although first generation DES reduced instent restenosis, still remained the unsolved problems such as stent thrombosis and restenosis in the era of DES. Second generation DES had been developed to improve the biocompatibility of stent coating focused on polymer compared to first generation DES, so that second generation stents showed better outcomes compared with first generation DES. On the other hands, in third generation DES, further refinement of DES involved more flexible stent platform. Promus ElementTM (Everolimus eluting stent, Boston Scientific, Nastick, MA) and Resolute Integrity® (Zotarolimus eluting stent, Medtronic Vascular, Santa Rosa, CA) are the third generation drug eluting stents which are designed to increase flexibility. In previous randomized controlled studies, both of these stents have shown at least non-inferior angiographic and clinical outcomes compared to second generation DES. However, there is lack of data about comparison of angiographic and clinical outcomes between Promus ElementTM and Resolute Integrity®.

IVUS is one of the widely used intracoronary imaging devices to provide more reproducible and accurate information about coronary anatomy than angiography in current practice.8 Optimal stent expansion assessed by intravascular ultrasound (IVUS) has been reported as an important factor to prevent stent thrombosis or restenosis.9 Accordingly, there have been many studies to evaluate the procedural or clinical benefit of IVUS guided angioplasty. However, The clinical benefit of IVUS-guided angioplasty with stent implantation is still in a controversy. In the previous studies, IVUS-guided stent implantation showed positive or negative beneficial effect on clinical outcomes according to their study subjects. However, the stents used in the previous studies are less useful in current practice of cardiology and there is lack of data of 3rd generation DES, which have different stent profiles and outcomes with their predecessors.

Thus we would perform a prospective randomized study in order to compare the efficacy of IVUS-guided angioplasty with conventional angioplasty-guided procedure in the long coronary lesion. Our main hypothesis is IVUS-guided 3rd generation DES implantation in the long coronary lesions would have better clinical outcomes compared with conventional angiography-guided strategy. We also intend to assess the clinical outcomes after Promus ElementTM and Resolute Integrity® implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Coronary artery disease and lesions which are candidate for treatment with drug eluting stent according to current clinical practice guidelines
* PCI for lesion(s) which needs a stent of 26mm or more
* Reference diameter from 2.25 to 4.0mm

Exclusion Criteria:

* Restenosis lesion
* Reference vessel diameter < 2.25 mm or > 4.0mm
* Primary PCI for STEMI
* Contraindication to anti-platelet agents
* Treated with any DES within 3 months at other vessel
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Life expectancy < 1 year

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2013-10; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of angiography or IVUS guided third generation stent implantation | 1 year after implantation
  MACEs including cardiovascular death, myocardial infarction, stent thrombosis, and target vessel revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea